CLINICAL TRIAL: NCT03789461
Title: An Open-label Pilot Study of Fecal Microbiota Transplant (FMT) to Induce Weight Loss in Obese Subjects
Brief Title: Fecal Microbiota Transplant (FMT) to Induce Weight Loss in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT-OB study
Record Dates: First submitted 2018-12-24; First posted 2018-12-28 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Obesity
Keywords: Fecal Microbiota Transplantation; FMT
MeSH Terms: conditions — Obesity | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): FMT infusion
  Interventions: Procedure: Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Fecal Microbiota Transplantation — FMT infusion (100-200ml) and Mucosal Microbiota Assessment (To assess the fecal and mucosal microbiota before and after FMT)

SUMMARY:
Obesity is associated with changes in the composition of the intestinal microbiota, and the obese microbiome appears to be more efficient in harvesting energy from the diet.

Fecal microbiota transplantation (FMT) represents a clinically feasible way to restore the gut microbial ecology, and has proven to be a breakthrough for the treatment of recurrent Clostridium difficile infection.

The therapy is generally well tolerated and appeared safe. No clinical studies have assessed the dosage of FMT in obese subjects.

DETAILED DESCRIPTION:
Recently, accumulating evidence supports a role of the enteric microbiota in the pathogenesis of obesity-related insulin resistance. Obesity is associated with changes in the composition of the intestinal microbiota, and the obese microbiome appears to be more efficient in harvesting energy from the diet. Colonization of germ-free mice with an 'obese microbiota' results in a significantly greater increase in total body fat than colonization with a 'lean microbiota', suggesting gut microbiota as an additional contributing factor to the pathophysiology of obesity. Obese and lean phenotypes can also be induced in germ-free mice by transfer of fecal microbiota from human donors. These data have led to the use of microbiota therapeutics as a potential treatment for metabolic syndrome and obesity.

Fecal microbiota transplantation (FMT) represents a clinically feasible way to restore the gut microbial ecology, and has proven to be a breakthrough for the treatment of recurrent Clostridium difficile infection. Furthermore, clinical trials are being conducted to evaluate its use for other conditions including inflammatory bowel disease, irritable bowel syndrome, diabetes mellitus, non-alcoholic steatohepatitis and hepatic encephalopathy. Early results in human have shown that FMT from lean donor when transplanted into subjects with metabolic syndrome resulted in a significant improvement in insulin sensitivity and an increased in intestinal microbial diversity, including a distinct increase in butyrate-producing bacterial strains. The therapy is generally well tolerated and appeared safe. No clinical studies have assessed the dosage of FMT in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75; and
2. BMI ≥28 kg/m^2 and < 45 kg/m^2; and
3. Written informed consent obtained

Exclusion Criteria:

1. Current pregnancy
2. Known history or concomitant significant gastrointestinal disorders (including Inflammatory Bowel Disease, current colorectal cancer)
3. Known history or concomitant significant food allergies
4. Immunosuppressed subjects
5. Known history of severe organ failure (including decompensated cirrhosis), kidney failure, epilepsy, acquired immunodeficiency syndrome
6. Current active sepsis
7. Known contraindications to oesophago-gastro-duodenoscopy (OGD)
8. Use of probiotic or antibiotics in recent 3 months
9. New drugs in the last three months that can impact on metabolism or body weight
10. Previous gastric or small intestinal surgery that alters gut anatomy such as fundoplication, gastric resection, gastric bypass, small bowel resection, ileoectomy, colectomy
11. Patients who have a confirmed current active malignancy or cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of at least 10% reduction in weight | 6 weeks
  Determine the proportion of at least 10% reduction in weight compared with baseline weight

SECONDARY OUTCOMES:
Proportion of subjects maintaining weight reduction | 12, 26, 52, 78, 104 weeks
  Proportion of subjects maintaining at least 10% reduction in weight compared with baseline
Proportion of subjects maintaining weight reduction | 6,12, 26, 52, 78, 104 weeks
  Proportion of subjects maintaining at least 5% reduction in weight compared with baseline
Changes in waist circumference | 6,12, 26, 52, 78, 104 weeks
  Changes in waist circumference compared with baseline
Decrease in waist to hip ratio and in total body weight | 6,12, 26, 52, 78, 104 weeks
  At least 5% decrease in waist to hip ratio and in total body weight
Change in biochemical parameters | 6 weeks
  Study samples will collected to characterize which microbiota favors FMT by performing metagenomics of gut microbiome in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Siew NG, Prof., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Turnbaugh PJ, Hamady M, Yatsunenko T, Cantarel BL, Duncan A, Ley RE, Sogin ML, Jones WJ, Roe BA, Affourtit JP, Egholm M, Henrissat B, Heath AC, Knight R, Gordon JI. A core gut microbiome in obese and lean twins. Nature. 2009 Jan 22;457(7228):480-4. doi: 10.1038/nature07540. Epub 2008 Nov 30. PMID 19043404
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Ridaura VK, Faith JJ, Rey FE, Cheng J, Duncan AE, Kau AL, Griffin NW, Lombard V, Henrissat B, Bain JR, Muehlbauer MJ, Ilkayeva O, Semenkovich CF, Funai K, Hayashi DK, Lyle BJ, Martini MC, Ursell LK, Clemente JC, Van Treuren W, Walters WA, Knight R, Newgard CB, Heath AC, Gordon JI. Gut microbiota from twins discordant for obesity modulate metabolism in mice. Science. 2013 Sep 6;341(6150):1241214. doi: 10.1126/science.1241214. PMID 24009397
- [Background] Smith MI, Yatsunenko T, Manary MJ, Trehan I, Mkakosya R, Cheng J, Kau AL, Rich SS, Concannon P, Mychaleckyj JC, Liu J, Houpt E, Li JV, Holmes E, Nicholson J, Knights D, Ursell LK, Knight R, Gordon JI. Gut microbiomes of Malawian twin pairs discordant for kwashiorkor. Science. 2013 Feb 1;339(6119):548-54. doi: 10.1126/science.1229000. Epub 2013 Jan 30. PMID 23363771
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Kassam Z, Lee CH, Yuan Y, Hunt RH. Fecal microbiota transplantation for Clostridium difficile infection: systematic review and meta-analysis. Am J Gastroenterol. 2013 Apr;108(4):500-8. doi: 10.1038/ajg.2013.59. Epub 2013 Mar 19. PMID 23511459
- [Background] Wong SK, Kong AP, Mui WL, So WY, Tsung BY, Yau PY, Chow FC, Ng EK. Laparoscopic bariatric surgery: a five-year review. Hong Kong Med J. 2009 Apr;15(2):100-9. PMID 19342735